CLINICAL TRIAL: NCT01795690
Title: Clinical Registry Describing Treatment Reality of Patients With Cancer-(Therapy)-Induced Anemia
Brief Title: Clinical Tumor Anemia Registry (TAR)
Acronym: TAR
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: ASORS (Arbeitsgemeinschaft Supportive Maßnahmen in der Onkologie, Rehabilitation und Sozialmedizin der Deutschen Krebsgesellschaft) (Unknown)
Responsible Party: Sponsor
Other Study IDs: iOM TAR
Record Dates: First submitted 2012-10-08; First posted 2013-02-21 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2014-12

CONDITIONS: Anemia
Keywords: Anemia; Cancer; Hemoglobin; Quality of Life; FACT-An; FACT-GP; Erythropoiesis-Stimulating Agents (ESA); Epoetin; Ferric Carboxymaltose; Blood Transfusions
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to record information of routine treatment of anemia in cancer patients in Germany. An overview of the current treatment of anemia in German outpatient centers and hospitals will be provided. Primary outcome parameters, e.g. improvement in hemoglobin levels and changes in QoL, as well as patient characteristics of different treatments will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant disease
* Hemoglobin level < 11 g/dl (female) or < 12 g/dl (male)
* Start of antianemic therapy no more than 7 days prior to informed consent
* Performance status 0 - 3 (Karnofsky-Index >= 40%)
* Minimum age: 18 years
* Informed written consent

Exclusion Criteria:

* Hypersensitivity against antianemic therapies
* Myelodysplastic Syndrome
* Experimental antianemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant diseases starting anti-anemic treatment
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Documentation of therapies | 12 weeks per patient
  Overview on the current routine treatment of anemia in cancer patients in Germany

SECONDARY OUTCOMES:
Change in hemoglobin levels and QoL | 12 weeks per patient
  Effectiveness of different antianemic treatments is investigated by measuring increase of hemoglobin levels and QoL (FACT-An and FACT-GP).
  Baseline in hemoglobin (before treatment) is compared with hemoglobin levels after treatment. Each patient is followed for a maximum of 12 weeks to obtain data about the course of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- iOMEDICO, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steinmetz T, Schroder J, Plath M, Link H, Vogt M, Frank M, Marschner N. Antianemic Treatment of Cancer Patients in German Routine Practice: Data from a Prospective Cohort Study-The Tumor Anemia Registry. Anemia. 2016;2016:8057650. doi: 10.1155/2016/8057650. Epub 2016 Feb 4. PMID 26966573